CLINICAL TRIAL: NCT06548581
Title: Radiographic and Patient Reported Outcomes Following Joint Arthrodesis Following the Use of the SpeedPlate™ Rapid Compression Implants: An Ambidirectional Cohort Study
Brief Title: The SpeedPlate™ Rapid Compression Implant Study (The SPRINT™ Study)
Acronym: SPRINT™
Status: Active, not recruiting | Type: Observational
Sponsor: Treace Medical Concepts, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP2024-1
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Joint Arthrodesis; Joint Fixation
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients who have had joint arthrodesis procedures using the SpeedPlate™ Rapid Compression Implants: Patients 14 years of age or older that have had MTP and/or TMT joint fixation with the SpeedPlate™ Rapid Compression Implants will be eligible to participate based on inclusion and exclusion criteria established in the study protocol.
  Interventions: Device: SpeedPlate™ Rapid Compression Implants

INTERVENTIONS:
Device: SpeedPlate™ Rapid Compression Implants — MTP and/or TMT joint fixation with SpeedPlate™ Rapid Compression Implants

SUMMARY:
Post-market, observational, multicenter, unblinded, ambidirectional cohort study to evaluate outcomes of study participants treated with the SpeedPlate™ product.

Up to 200 participants will be treated in this study at (up to) 15 clinical sites.

Patients 14 years of age or older that have had MTP and/or TMT joint fixation with the SpeedPlate™ Rapid Compression Implants will be eligible to participate based on the inclusion and exclusion criteria defined in this protocol.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate:

1. Healing/union rates following joint fixation using the SpeedPlate™ Rapid Compression Implants
2. Whether early weight-bearing (WB) following joint fixation using the SpeedPlate™ Rapid Compression Implants affects the healing/union rates
3. Quality of life, pain scores and patient satisfaction following joint arthrodesis using the SpeedPlate™ Rapid Compression Implants

ELIGIBILITY:
Inclusion Criteria:

Patients satisfying the following criteria will be considered and eligible for participation:

1. Patients who have had MTP and/or TMT joint fixation using at least one SpeedPlate™ Rapid Compression Implant (Index Procedure);
2. Males and females ages 14 years of age or older at the time of the Index Procedure;
3. Patients who have completed at least their 6-week post-operative visit but have not yet completed their 12-month post-operative visit;
4. Adequate pre-operative AP and lateral weight-bearing radiographs collected within 6 months of the Index Procedure;
5. Patients must be capable of completing self-administered questionnaires;
6. Willing and able to provide written informed consent.

Exclusion Criteria:

Patients satisfying the following criteria will not be eligible for participation:

1. Female patients of childbearing potential with positive pregnancy result at time of consent;
2. Unwilling or unable to schedule and return for follow-up visits;
3. Surgery for MTP or TMT joint arthrodesis on operative foot prior to Index Procedure;
4. Joint arthrodesis using other plating constructs in addition to the SpeedPlate™ Implant(s) at MTP or TMT joint at the time of Index Procedure;
5. Surgeries on operative foot involving fusion of the foot or ankle joints prior to, or at the time of, Index Procedure (other than hammertoe or lesser toes/digits);
6. Clinically significant neuropathy at time of Index Procedure;
7. Untreated Moderate - Severe Osteoarthritis of 1st, 2nd, or 3rd TMT or MTP during the Index Procedure;
8. Untreated Moderate - Severe Osteoarthritis of the foot or ankle outside of the 1st, 2nd or 3rd TMT or MTP joints at the time of Index Procedure;
9. BMI >40 kg/m² at time of Index Procedure;
10. Use of structural bone graft during the Index Procedure;
11. Additional concomitant procedure during the Index Procedure that would have altered patient's ability to early weight-bear post-procedure.
12. Patient is actively involved with a workman's compensation case or is currently involved in litigation;
13. Patient is currently or has participated in a clinical study in the last 30 days prior to signing informed consent or is considering participation in another research protocol during this study; exceptions to this include survey clinical studies with no treatment or if participant is greater than 12 months post-procedure in either the Treace ALIGN3D™, Mini3D™ or MTA3D™ study without ongoing protocol defined adverse events;
14. Patient has a condition or finding that, in the opinion of the Investigator, may jeopardize the patient's well-being, the soundness of this clinical study, or could interfere with provision of informed consent, completion of tests, therapy, or follow-up.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients 14 years of age or older that have had MTP and/or TMT joint fixation with the SpeedPlate™ Rapid Compression Implants.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate union vs non-union | 12 Months
  Evaluate clinical/radiographic healing (union vs non-unio). Non-union is defined as radiographic lucency and clinical pain at the 1st, 2nd, and/or 3rd TMT or MTP joint at 12 months post Index.

SECONDARY OUTCOMES:
Evaluate the Intermetatarsal Angle | 6 Weeks, 3-4 Months, 6 Months, 12 Months, 24 Months
  Evaluate change in radiographic angular/positional alignment of the Intermetatarsal Angle - (IMA) before and after Index.
Evaluate the Hallux Valgus Angle | 6 Weeks, 3-4 Months, 6 Months, 12 Months, 24 Months
  Evaluate change in radiographic angular/positional alignment of the Hallux Valgus Angle (HVA) before and after Index.
Evaluate the Tibial Sesamoid | 6 Weeks, 3-4 Months, 6 Months, 12 Months, 24 Months
  Evaluate change in radiographic angular/positional alignment of the Tibial Sesamoid Position (TSP) before and after Index.
Evaluate time to start weight-bearing in a boot. | Days after surgery - on average up to 2 weeks
  Time to start of weight-bearing in boot, in days.
Evaluate time to start weight-bearing in shoes. | Days after surgery - on average up to 6 weeks
  Time to start of weight-bearing in shoes, in days.
Evaluate time to start unrestricted activity. | Days after surgery - on average up to 4 months
  Time to return to full unrestricted activity, in days.
Evaluate patient-reported pain, post surgery. | 6 Months, 12 Months, 24 Months
  Reported pain via Visual Analog Scale (VAS) at 6-, 12- and 24-months post-procedure. The VAS pain scale is measured from 0-10 with 0 being "pain free" to 10 being "unconscious - pain makes you pass out".
Evaluate patient-reported quality of life, post surgery. | 6 Months, 12 Months, 24 Months
  Quality of Life (Manchester-Oxford Foot Questionnaire) defined as the total domain score measured at 6-, 12- and 24-months post-procedure. The MOxFQ is a series of 16 quality of life questions related to a patient's foot - from pain, appearance, and functionality. Answers range from "none of the time to all of the time", "none to severe" and "no nights to every night".
Evaluate patient-reported satisfaction, post surgery. | 12 Months, 24 Months
  Post-Operative Patient Satisfaction at 12- and 24-months post-procedure. The Post-Op Patient Satisfaction questionnaire asks a series of 10 quality of life questions related to the patient's surgical and recovery experience as related to: pain, function, foot alignment, and foot aesthetics. The answers range mostly from "better, worse, same" and "satisfied, unsatisfied".
Evaluate non-surgical clinical complications or health conditions that could affect outcomes related to the implants or procedure. | 24 Months
  Percentage of participants experiencing at least one clinical complication related to the SpeedPlate™ Rapid Compression Implants, to the joint arthrodesis procedure, or to other health conditions that could affect outcome measures and not requiring surgical intervention through the 24-month post-operative visit.
Evaluate surgical clinical complications or health conditions that could affect outcomes related to the implants or procedure. | 24 Months
  Percentage of participants experiencing at least one clinical complication related to the SpeedPlate™ Rapid Compression Implants, to the joint arthrodesis procedure, or to other health conditions that could affect outcome measures through the 24-month post-operative visit and requiring one or more of the following subsequent secondary surgical interventions (SSSI):
  1. hardware removal (any reason, hardware not replaced)
  2. revision of bone for delayed union or non-union (e.g. bone graft)
  3. hardware failure (e.g. broken hardware) requiring supplemental fixation or hardware replacement
  4. wound healing (hardware not replaced or removed)
  5. infection at the surgical site (hardware not replaced or removed)
  6. other complication requiring surgical intervention

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Decatur Orthopaedic Clinic, Decatur, Alabama
  - Orlando Foot and Ankle Clinic, Orlando, Florida
  - JCMG - Podiatry, Jefferson City, Missouri
  - Ohio Foot and Ankle Center, Stow, Ohio
  - Foot and Ankle Associates of North Texas, Keller, Texas